CLINICAL TRIAL: NCT04642144
Title: Effect of Infusion of Yerba Mate (Ilex Paraguariensis) Associated or Not With Carbohydrate Intake on Oxidative Stress, Pshysiological and Performance Parameters of Trained Cyclists
Brief Title: Effect of Infusion of Yerba Mate on Oxidative Stress, Physiology, and Performance of Trained Cyclists
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Santa Catarina (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Principal Investigator, Brunna Cristina Bremer Boaventura, Clinical Professor, Universidade Federal de Santa Catarina
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 04545218.1.0000.0121
Record Dates: First submitted 2020-11-06; First posted 2020-11-24 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-03

CONDITIONS: Sports Performance; Sports Nutritional Sciences; Endurance Performance
Keywords: Ilex paraguariensis; Yerba mate; Cycling; Ergogenic aids; Metabolism; Plant-based; Nutrition

STUDY DESIGN:
Intervention Model Description: A group with yerba mate infusion and carbohydrate meal, a group with only yerba mate infusion, and a group with water and carbohydrate. The washout period between treatments will be seven days
Masking Description: Not Masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Yerba mate and carbohydrate (Experimental): Consumption of yerba mate infusion and carbohydrate-based meal.
  Interventions: Other: Yerba mate infusion; Other: Carbohydrate meal
- Yerba mate and fasting (Active Comparator): Consumption of yerba mate infusion and stay in a fasting state.
  Interventions: Other: Yerba mate infusion
- Carbohydrate and water (Active Comparator): Carbohydrate meal consumption and water intake.
  Interventions: Other: Carbohydrate meal

INTERVENTIONS:
Other: Yerba mate infusion — Yerba mate infusion intervention is characterized by the consumption of the infusion of yerba mate for 7 days preceding the test, with consumption of the infusion right before the exercise protocol test, without consumption of a carbohydrate-based meal, keeping the individual fasted.
  Yerba mate and carbohydrate intervention is characterized by the consumption of the infusion of yerba mate for 7 days preceding the test, with consumption of a meal based on carbohydrate right before the exercise protocol test with another infusion of yerba mate.
  Arms: Yerba mate and carbohydrate; Yerba mate and fasting
Other: Carbohydrate meal — Carbohydrate meal intervention is characterized by the consumption of a carbohydrate-based meal right before the exercise protocol test, without consumption yerba mate infusion.
  Arms: Carbohydrate and water; Yerba mate and carbohydrate

SUMMARY:
This project comes forward with investigations regarding the use of yerba mate infusion in sports performance, providing new knowledge about the effects of its consumption on the performance of trained individuals, thus elucidating new mechanisms of ergogenic action of the plant in characteristics of dietary management indicated for trained individuals, besides investigating on the action of the bioactive compounds of the plant in the metabolism and performance of athletes and the physiological aspects.

DETAILED DESCRIPTION:
In this study, participants will be randomized into three groups: a group with yerba mate infusion and carbohydrate meal, a group with only yerba mate infusion, and a group with water and carbohydrate. The washout period between treatments will be seven days. The experimental protocol will be carried out in the same period of the day (± 3h) to minimize the interference of biological variations.

Before starting the procedures for data collection, the individuals invited to participate in the study will be informed about the objectives and methods of the research and then, if accepted, they will sign the informed consent form. The study will be divided into four stages (baseline and the three different interventions). The baseline period comprises two meetings, the first of which is to carry out a questionnaire to identify the participant, to carry out blood collection of the intermediate vein of the arm, to make the analysis of body composition and to be instructed on the exercise and feeding procedures during the experimental protocol. In the second meeting of the baseline period, the participants will be submitted to an incremental protocol on the cycle ergometer, and the data from this test will be used for the application of the experimental exercise protocol performed later with dietary interventions. From the incremental test, the maximum aerobic power, peak oxygen volume, maximum heart rate, and lactate thresholds, energy substrate consumption, and perceived exertion will be determined. In the three visits following the baseline period, according to randomization, interventions will be carried out with the infusion of yerba mate and carbohydrate meal, with only the infusion of yerba mate and with water and carbohydrate meal. In intervention groups with yerba mate infusion, participants will be asked to ingest seven days before the exercise protocol the same amount of yerba mate infusion as the test day (250 mL). In this way, individual packages of ultra-refined yerba mate containing 5 g, the necessary materials, and guidelines for the proper preparation of the infusion will be provided. In groups that receive the carbohydrate meal, participants will be offered, one hour before starting the exercise protocol, white bread with corn syrup, which will be adjusted to their individual carbohydrate needs, in quantities that make up a total of 1g of carbohydrate per kg of bodyweight of the participant, as recommended by the American College of Sports Medicine and the Academy of Nutrition and Dietetics, Dietitians of Canada.

In all visits, participants will be instructed to arrive at the physical effort laboratory of the Federal University of Santa Catarina in a 10-hour overnight fast, following the protocols of dietary control and physical exercise in which they must maintain their usual pattern of exercises and food throughout the study, except for the restriction of the consumption of micronutrient food supplements, beverages with antioxidant and stimulating properties already known, such as green tea, black tea, and wines, which may interfere with the results of the study due to the similarity of bioactive compounds from yerba mate in the composition of these drinks. In all these visits in which there will be dietary intervention, the participants will assess their body composition and perform the exercise protocol to assess their performance.

In each of the three intervention visits, 60 minutes before the exercise protocol, a carbohydrate meal will be offered (for when the individual is randomized to the group in which this meal is consumed); 40 minutes before the exercise protocol, the infusion of yerba mate or water (250 mL) will be performed; immediately before the exercise protocol, blood will be collected from the intermediate vein of the arm to observe the increase in phenolics in the blood promoted by the ingestion of the yerba mate infusion. Soon after, it will be the realization of the effective exercise protocol to measure performance. During the execution of the exercise protocol, blood samples will be collected from the earlobe to check the variations of lactate and glucose. At the end of the exercise protocol, a new blood collection will be performed in the middle vein of the arm to assess biochemical variations that may have been influenced after exercise.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Age between 20 and 45 years
* Minimum of two years of experience with training and competitions

Exclusion Criteria:

* Individuals who present clinical condition of disease
* Smokers
* Continuous use of medications and/or dietary supplements
* Show aversion, intolerance, or complications resulting from ingesting the YERBA MATE infusion or any of its components

Ages: 25 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2021-01-05 (Actual); Study Completion 2021-01-21 (Actual)

PRIMARY OUTCOMES:
Power (kilojoules) | Pre and post test on cycle ergometer, through study completion, an average of 1 month.
  To analyze the effects of the infusion of yerba mate drink on potency.

SECONDARY OUTCOMES:
Oxygen Consumption (% VO2 max) | During cycle ergometer test, through study completion, an average of 1 month.
  To determine and compare the physiological responses regarding oxygen consumption with yerba mate consumption.

OTHER OUTCOMES:
Total Antioxidant Capacity (mmol/L) | Pre and post test on cycle ergometer, through study completion, an average of 1 month.
  To measure the total antioxidant capacity before and after exercise after drinking yerba mate infusion.
Total Phenolic Compounds Content (ug/mL) | Pre and pos intake of yerba mate infusion, through study completion, an average of 1 month.
  To determine the total phenolic compounds content on blood after drinking yerba mate.

CONTACTS AND LOCATIONS:
Overall Officials: Brunna Boaventura, PhD, Principal Investigator — Federal University of Santa Catarina
Locations (1):
- Department of Nutrition, Florianópolis, Santa Catarina, Brazil

IPD SHARING:
Plan to Share IPD: No
Individuals' data are limited to the creation of results only for the research that our group is proposing to develop, not considering the sharing of individual data, keeping them confidential.

REFERENCES:
- [Derived] Krolikowski TC, Borszcz FK, Panza VP, Bevilacqua LM, Nichele S, da Silva EL, Amboni RDMC, Guglielmo LGA, Phillips SM, de Lucas RD, Boaventura BCB. The Impact of Pre-Exercise Carbohydrate Meal on the Effects of Yerba Mate Drink on Metabolism, Performance, and Antioxidant Status in Trained Male Cyclists. Sports Med Open. 2022 Jul 16;8(1):93. doi: 10.1186/s40798-022-00482-3. PMID 35841429